CLINICAL TRIAL: NCT04185974
Title: Carbon Ion Re-Radiotherapy in Patients With Recurrent or Progressive Locally Advanced Head-and-Neck Cancer: A Phase-II Study to Evaluate Toxicity and Efficacy
Brief Title: Carbon Ion Re-Radiotherapy in Patients With Recurrent or Progressive Locally Advanced Head-and-Neck Cancer
Acronym: CARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Head of department, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADONK-CARE-2018
Record Dates: First submitted 2019-11-25; First posted 2019-12-04 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Head-and-Neck Cancer

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C12 irradiation (Experimental): Evaluation of Safety and Toxicity of C12 ion reirradiation
  Interventions: Radiation: C12 re-irradiation
- Photon irradiation (Active Comparator): Evaluation of Safety and Toxicity of photon re-irradiation
  Interventions: Radiation: Photon re-irradiation

INTERVENTIONS:
Radiation: C12 re-irradiation — 51 Gy(RBE) or 54 Gy
  Arms: C12 irradiation
Radiation: Photon re-irradiation — 54 Gy(RBE) or 60 Gy
  Arms: Photon irradiation

SUMMARY:
After multimodal therapy of head-and-neck tumors, patients often develop local recurrence, locally progressive disease or second primary tumors. In this highly pre-treated patient cohort, therapeutic options are limited. Patients that are not candidates for salvage surgery may benefit from re-irradiation. Despite recent technical advances, re-irradiation is associated with severe side effects. Carbon ion Re-Radiotherapy (reCIRT) has shown encouraging results in retrospective analyses with moderate toxicity.

In the current Phase-II CARE-trial, reCIRT and conventional photon re-irradiation in patients with recurrent or progressive locally advanced head-and-neck cancer will be assessed regarding toxicity/ safety, local progression-free survival, overall survival and quality-of-life.

DETAILED DESCRIPTION:
The incidence of head-and-neck cancer worldwide amounts to around 550.000 cases per year, with male patients affected significantly more often. Common risk factors are smoking, alcohol, viral infections, immunodeficiency or genetic factors. Locally advanced head-and-neck tumors can lead to severe symptoms such as dysphagia, cachexia and tumor pain with a significant decrease of the quality-of-life. The prognosis depends on multiple factors such as TNM-staging, tumor volume, histology, general condition, age and smoking. Further risk factors are positive resection margins, extracapsular extension and perineural invasion. While metastatic spread significantly decreases overall survival, the life-limiting problem in patients with head-and-neck cancer is locally invasive and destructive tumor growth leading to a decrease of the performance status and quality of life. After multimodal therapy of locally advanced head-and-neck tumors, around 30 - 50% of patients will develop local recurrence or locally progressive disease and up to 8% of patients with HNSCC will develop a second primary tumor in the head-and-neck .

ELIGIBILITY:
Inclusion Criteria:

* Locally recurrent / progressive head-and-neck cancer after initial radiation therapy
* Microscopic or macroscopic tumor after salvage surgery
* Indication for re-irradiation
* Completed wound healing after surgical intervention
* Karnofsky-Performance-Score ≥ 60
* Age ≥ 18 years
* Written informed consent (must be available before enrolment in the trial)
* Ability of subject to understand character and individual consequences of the trial
* For women with childbearing potential, (and men) adequate contraception
* Submission of previous radiotherapy records

Exclusion Criteria:

* Re-irradiation of malignancy in the larynx
* Diagnosed plasmocytoma, sarcoma or chordoma
* Previous re-irradiation in-field
* Time interval < 6 months after initial radiotherapy
* Distant metastases (except pulmonary metastases)
* Patients who have not recovered from acute toxicities of prior therapies
* Refusal of the patients to take part in the study
* Pregnant or lactating women
* Known carcinoma <5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* Participation in another clinical study or observation period of competing trials, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
safety of carbon ion re-irradiation | 6 month
  the rate of patients with an acute/subacute toxicity CTCAE v5.0 ≥ grade 3
toxicity of carbon ion re-irradiation | 6 month
  the rate of patients with an acute/subacute toxicity CTCAE v5.0 ≥ grade 3

SECONDARY OUTCOMES:
progression-free survival | 12 month
  Local progression-free survival
Overall survival | 12 month
  within 12 month after re-irradiation
Score on EORTC QLQ C30 Quality of life questionaire | within 12 month after re-irradiation
  EORTC (European Organization for Research and. Treatment of Cancer) QLQ (quality of life questionnaire) C30, score 1-6, high score means worse outcome
Score on EORTC QLQ H&N35 Quality of life questionaire | within 12 month after re-irradiation
  QLQ (quality of life questionnaire)-H&N (Head and neck) 35, score 1-6, high score means worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Held T, Lang K, Regnery S, Weusthof K, Hommertgen A, Jakel C, Tonndorf-Martini E, Krisam J, Plinkert P, Zaoui K, Freudlsperger C, Moratin J, Krauss J, Harrabi SB, Herfarth K, Debus J, Adeberg S. Carbon ion reirradiation compared to intensity-modulated re-radiotherapy for recurrent head and neck cancer (CARE): a randomized controlled trial. Radiat Oncol. 2020 Aug 5;15(1):190. doi: 10.1186/s13014-020-01625-0. PMID 32758267